CLINICAL TRIAL: NCT01648920
Title: A Study to Explore the Utility of Fractional Exhaled Nitric Oxide (FeNO) Compared With Methacholine Challenge (MCC) Testing in the Assessment of Patients With Suspected But Undiagnosed Asthma
Status: Completed | Type: Observational
Sponsor: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: AER-044
Record Dates: First submitted 2012-07-05; First posted 2012-07-25 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Asthma
Keywords: Asthma; Suspected but undiagnosed asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FeNO: Participants with suspected but undiagnosed asthma will have a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit. Following that they will have a Methacholine Challenge (MCC) test performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests
  Interventions: Device: NIOX MINO® Instrument (09-1100)

INTERVENTIONS:
Device: NIOX MINO® Instrument (09-1100) — The NIOX MINO® Instrument (09-1100) is a 10 second test based on exhaled breath measured at a 50 ml/second flow rate.

SUMMARY:
Objective: To explore the utility of Fractional Exhaled Nitric Oxide (FeNO) compared with Methacholine Challenge (MCC) testing in assessing patients with suspected but undiagnosed asthma

Number of participants: Approximately 50 subjects will be enrolled

Reference product: NIOX MINO® Instrument (09-1100)

Performance assessments: FeNO measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual. MCC testing will be performed according to the ATS guidelines and the allergy and asthma specialists procedure for conducting MCC tests

Safety assessments: The Investigator is responsible for the detection, reporting, and documentation of events meeting the definition of an Adverse Event (AE) and/or Serious Injuries as provided in this clinical investigation plan from the time that informed consent has been provided and during the study period

Criteria for evaluations: This is an exploratory study and there are currently no plans for a formal statistical analysis. Information gained from this study may used to design and power subsequent studies in patients with suspected but undiagnosed asthma. Information collected will be summarized in a clinical study report

DETAILED DESCRIPTION:
INTRODUCTION

Overview:

The measurement of exhaled nitric oxide (FeNO) is the only clinical test for measuring airway inflammation that can be performed consistently and accurately in clinical practice at the point-of-care. Airway inflammation is now recognized as the central mechanism in the pathogenesis of asthma. The measurement of FeNO with the NIOX MINO® device provides a rapid, noninvasive, and inexpensive tool to assess airway inflammation in inflammatory airway diseases such as asthma. The test is easy to perform and requires minimal training for the operator to conduct the test.

Role of Exhaled Nitric Oxide (FeNO):

FeNO has evolved as a predictive and prognostic biomarker for airway inflammation. Nitric oxide (NO) gas is produced in the epithelial cells of the bronchial wall as an intrinsic part of the inflammatory process.

Measuring the amount of FeNO is useful in the initial assessment of patients with chronic cough or non-specific respiratory symptoms suggestive of asthma, and for the management of patients with established asthma who are receiving corticosteroid treatment.

Intended Use:

NIOX MINO® measures Nitric Oxide (NO) in human breath. Nitric Oxide is frequently increased in inflammatory processes such as asthma. The fractional NO concentration in expired breath (FeNO) can be measured by NIOX MINO® with assurance that such measurements are repeatable and according to guidelines for NO measurement established by the American Thoracic Society.

Rationale for Study:

The burden of asthma in the U.S. is significant and growing. In addition, it has been established that asthma is both over- and under- diagnosed. Equally concerning is the fact that nearly 75% of these misdiagnosed patients are receiving anti-asthma treatments. Data such as these point out the need for a simple, inexpensive and reliable way to establish the diagnosis of asthma.

Presently, the assessment of patients with suspected but undiagnosed asthma is to perform Methacholine Challenge (MCC) testing to evaluate airway hyperresponsiveness. However, MCC, testing is difficult, time-consuming, and costly and also involves some level of risk to the patient. Nonetheless, there is some evidence that FeNO testing may be able to identify the patients who actually have asthma among those with suspected but undiagnosed asthma who have normal pulmonary function tests, thus potentially eliminating the need for MCC testing in many patients.

CLINICAL INVESTIGATION OBJECTIVES To explore the utility of FeNO compared with MCC in assessing patients with suspected but undiagnosed asthma.

CLINICAL INVESTIGATION PLAN

This is an exploratory, multi-center, single-visit, outpatient study. Approximately 50 subjects will participate in the study during an (approximately 8-16 week study enrollment period:

* Demographics
* Physical Characteristics
* Smoking history (cigarettes only)
* FeNO
* Spirometry
* Asthma and Allergy Specialists MCC Test Procedure

Subject discharge from the study:

Once all information has been collected and all procedures have been performed, the subject will be discharged from the clinic and their study participation will be complete

Medical device:

The NIOX MINO® was initially cleared by the FDA on March 4, 2008 as a new hand-held device for the measurement of exhaled Nitric Oxide, a marker of eosinophilic airway inflammation. The most recent clearance by the FDA was on September 2, 2010 for Instrument (09-1100), which will be used in this study. NIOX MINO® can be used in children 7-17 years of age and in adults 18 years of age or older in the initial assessment and management of asthma.

The NIOX MINO® is a 10 second test based on exhaled breath measured at a 50 ml/second flow rate. Results are provided at the point of care within 2 minutes after the successful completion of the breath test. The test cannot be influenced by patient effort or variations in the clinician's test technique.

Definitions:

Adverse event: Any incident where the use of a medical device (including in vitro diagnostics) is suspected to have resulted in an adverse outcome in a patient.

Serious Injury means injury or illness that:

* Is life-threatening
* Results in permanent impairment of a body function or permanent damage to a body structure, or
* Necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.

Malfunction: the failure of a device to meet its performance specifications or otherwise perform as intended.

Caused or contributed: the death or serous injury was or may have been attributed to a medical device, or that the medical device was or may have been a factor in a death or serious injury, including events occurring as a result of:

* Failure
* Malfunction
* Improper or inadequate design
* Manufacture
* Labeling
* User error

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected but undiagnosed asthma that are scheduled to undergo MCC testing as part of the routine evaluation of suspected asthma.

Exclusion Criteria:

* Concurrent Conditions or Disease:
* current diagnosis of asthma, COPD, or other chronic respiratory disease
* upper or lower respiratory infection (including the common cold) that has not resolved within 4 weeks prior to the MCC test

Medication Use:

* scheduled use of asthma and allergy medication(s) should be discontinued at least 48 hours prior to MCC testing
* rescue medications should be discontinued at least 8 hour prior to MCC testing

Smoking:

- smoking should be avoided for at least 8 hours prior to MCC testing

Exercise:

- exercise or outdoor activity should be avoided for at least 2 hours prior to testing

Vaccinations:

-vaccinations should be avoided at least 2 weeks prior to MCC testing

Study participation outside of the protocol:

-subjects currently enrolled in studies of investigational or non-investigational drugs or medical devices and/or who participated in these studies within 30 days prior to this study are excluded

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects, approximately 7 years of age and above with suspected but undiagnosed asthma that are scheduled to undergo Methacholine Challenge (MCC) testing as part of the routine evaluation of suspected asthma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Anolik, MD, Principal Investigator — Allergy and Asthma Specialists, PC
Locations (8):
- United States (8):
  - Allergy and Asthma Specialists, PC, Blue Bell, Pennsylvania
  - Allergy and Asthma Specialists, PC, Collegeville, Pennsylvania
  - Allergy and Asthma Specialists, PC, Doylestown, Pennsylvania
  - Allergy and Asthma Specialists, PC, Jenkintown, Pennsylvania
  - Allergy and Asthma Specialists, PC, King of Prussia, Pennsylvania
  - Allergy and Asthma Specialists, PC, Lansdale, Pennsylvania
  - Allergy and Asthma Specialists, PC, Philadelphia, Pennsylvania
  - Allergy and Asthma Specialists, PC, Pottsville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- FeNO: Participants with suspected but undiagnosed asthma had a fractional exhaled nitric oxide (FeNO) measurement taken by NIOX MINO® Instrument (09-1100) according to the 'Perform FeNO Measurement' guidelines on page 7 of the NIOX MINO® User Manual (February 2011) during their study visit. Following that they had a Methacholine Challenge (MCC) test performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests
  NIOX MINO® Instrument (09-1100): The NIOX MINO® Instrument (09-1100) is a 10 second test based on exhaled breath measured at a 50 ml/second flow rate.
Period: Overall Study
Arm/Group | FeNO
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 50 subjects appeared to be a representative sample to generate summary statistics to characterize the data collected.
Arm/Group | FeNO
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 24.7 [7 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Methacholine Challenge (MCC) Results
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests will be performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 50
participants
  >= 20% decrease in FEV1 from BL MCC Dilution | 14
  <20% Decrease in FEV1 from BL MCC Dilution | 36

2. Primary Outcome: Mean FeNO Levels by Methacholine Challenge (MCC) Results: MCC Results
Description: as for outcome 1
Time Frame: approximately 1-hour
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | FeNO
Number analyzed (Participants) | 50
parts per billion (ppb)
  >= 20% decrease in FEV1 from BL MCC Dilution | 17.4 (12.54)
  <20% Decrease in FEV1 from BL MCC Dilution | 17.7 (9.77)

3. Primary Outcome: FeNO by Methacholine Challenge (MCC) Results: FeNO <25ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements will be performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests will be performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. A positive response to methacholine challenge is defined as a greater than or equal to 20% decrease in FEV1 at a methacholine dose less than or equal to 16mg/ml from baseline in response to methacholine. A negative response to methacholine challenge is defined as a less than 20% decrease in FEV1 at a methacholine dose less than or equal to 16mg/ml from baseline.
Time Frame: approximately 1-hour
Population: Participants with a FeNO < 25 ppb
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 38
participants
  Positive Response to MCC | 12
  Negative Response to MCC | 26

4. Primary Outcome: FeNO by Methacholine Challenge (MCC) Results: FeNO >=25ppb to <=50ppb
Description: as for outcome 3
Time Frame: approximately 1-hour
Population: Participants with FeNO >= 25 ppb to <= 50 ppb
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 11
participants
  Positive Response to MCC | 1
  Negative Response to MCC | 10

5. Primary Outcome: FeNO by Methacholine Challenge (MCC) Results: FeNO >50ppb
Description: as for outcome 3
Time Frame: approximately 1-hour
Population: Participants with FeNO >50ppb
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 1
participants
  Positive Response to MCC | 1
  Negative Response to MCC | 0

6. Primary Outcome: Asthma Diagnosis by MCC Results: Positive MCC Response
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements was performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. A positive response to methacholine challenge is defined as a greater than or equal to 20% decrease in FEV1 at a methacholine dose less than or equal to 16mg/ml from baseline in response to methacholine.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 14
participants
  Asthma | 11
  Non-Asthma | 3

7. Primary Outcome: Asthma Diagnosis by MCC Results: Negative MCC Response
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements was performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. A negative response to methacholine challenge is defined as a less than 20% decrease in FEV1 at a methacholine dose less than or equal to 16mg/ml from baseline.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 36
participants
  Asthma | 0
  Non-Asthma | 36

8. Primary Outcome: Asthma Diagnosis by FeNO: FeNO <25ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 38
participants
  Asthma | 10
  Non-Asthma | 28

9. Primary Outcome: Asthma Diagnosis by FeNO: FeNO >=25ppb to <= 50ppb
Description: as for outcome 8
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 11
participants
  Asthma | 0
  Non-Asthma | 11

10. Primary Outcome: Asthma Diagnosis by FeNO: FeNO >50ppb
Description: as for outcome 8
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 1
participants
  Asthma | 1
  Non-Asthma | 0

11. Primary Outcome: Asthma Diagnosis by FeNO: Mean FeNO Value
Description: as for outcome 8
Time Frame: approximately 1-hour
Measure: Mean (Standard Deviation); unit: Parts per billion (ppb)
Arm/Group | FeNO
Number analyzed (Participants) | 50
Parts per billion (ppb)
  Asthma | 16.9 (12.21)
  Non-Asthma | 17.8 (10.11)

12. Primary Outcome: Sensitivity (%) for FeNO
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. Sensitivity is a way of saying how likely a test is positive if you have a disease and is expressed as (%) percent. For this study, sensitivity was the ability of FeNO to correctly identify a study participant who has asthma.
Time Frame: approximately 1-hour
Measure: Number; unit: percent
Arm/Group | FeNO
Number analyzed (Participants) | 50
percent
  FeNO <= 10 ppb | 35.7
  FeNO <= 15 ppb | 57.1
  FeNO <=20 ppb | 85.7
  FeNO <=25 ppb | 85.7
  FeNO <=30 ppb | 85.7
  FeNO <= 35 ppb | 85.7
  FeNO <= 40 ppb | 92.9
  FeNO <= 45 ppb | 92.9
  FeNO <= 50 ppb | 92.9
  FeNO <= 55 ppb | 100.0

13. Primary Outcome: Specificity (%) for FeNO
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. Specificity is a way of saying how likely a test is negative if you do not have a disease and is expressed as (%) percent. For this study, specificity was the ability of FeNO to correctly identify a study participant who does not have asthma.
Time Frame: approximately 1-hour
Measure: Number; unit: percent
Arm/Group | FeNO
Number analyzed (Participants) | 50
percent
  FeNO <= 10 ppb | 75.0
  FeNO <= 15 ppb | 55.6
  FeNO <=20 ppb | 33.3
  FeNO <=25 ppb | 25.0
  FeNO <=30 ppb | 11.1
  FeNO <= 35 ppb | 2.8
  FeNO <= 40 ppb | 2.8
  FeNO <= 45 ppb | 0.0
  FeNO <= 50 ppb | 0.0
  FeNO <= 55 ppb | 0.0

14. Primary Outcome: Positive Predictive Value (%) for FeNO
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. Positive predictive value is a way of saying the likelihood a positive test means you have a disease. In this study, it is defined as the percentage of study participants with a high FeNO who have asthma.
Time Frame: approximately 1-hour
Measure: Number; unit: percent
Arm/Group | FeNO
Number analyzed (Participants) | 50
percent
  FeNO <= 10 ppb | 35.7
  FeNO <= 15 ppb | 33.3
  FeNO <=20 ppb | 33.3
  FeNO <=25 ppb | 30.8
  FeNO <=30 ppb | 27.3
  FeNO <= 35 ppb | 25.5
  FeNO <= 40 ppb | 27.1
  FeNO <= 45 ppb | 26.5
  FeNO <= 50 ppb | 26.5
  FeNO <= 55 ppb | 28.0

15. Primary Outcome: Negative Predictive Value (%) for FeNO
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests will be compared against final asthma diagnosis. Negative predictive value is a way of saying the likelihood of a negative test means you do not have disease. In this study it is defined as the percentage of study participants with a low FeNO who do not have asthma.
Time Frame: approximately 1-hour
Measure: Number; unit: percent
Arm/Group | FeNO
Number analyzed (Participants) | 50
percent
  FeNO <= 10 ppb | 75.0
  FeNO <= 15 ppb | 76.9
  FeNO <=20 ppb | 85.7
  FeNO <=25 ppb | 81.8
  FeNO <=30 ppb | 66.7
  FeNO <= 35 ppb | 33.3
  FeNO <= 40 ppb | 50.0

16. Primary Outcome: FeNO Values by ICS Use: FeNO <25ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests were compared against final asthma diagnosis. Data are presented for participants with FeNO <25ppb who either did not use Inhaled Corticosteroids (ICS) or did use Inhaled Corticosteroids.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 38
participants
  No ICS Use | 34
  Yes ICS Use | 4

17. Primary Outcome: FeNO Values by ICS Use: FeNO >= 50ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests were compared against final asthma diagnosis. Data are presented for participants with FeNO >=50ppb who either did not use Inhaled Corticosteroids (ICS) or did use Inhaled Corticosteroids.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 1
participants
  No ICS Use | 1
  Yes ICS Use | 0

18. Primary Outcome: FeNO Values by ICS Use: FeNO >= 25ppb to <= 50ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests were compared against final asthma diagnosis. Data are presented for participants with FeNO <=25ppb to <=50ppb who either did not use Inhaled Corticosteroids (ICS) or did use Inhaled Corticosteroids.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 11
participants
  No ICS Use | 10
  Yes ICS Use | 1

19. Primary Outcome: FeNO Values by Smoking Status: FeNO <25ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests were compared against final asthma diagnosis. Data are presented for participants with FeNO <25ppb who either did not smoke previously or are current smokers.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 38
participants
  No Previous Smoker | 34
  Current Smoker | 4

20. Primary Outcome: FeNO Values by Smoking Status: FeNO >= 25ppb to <= 50ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests were compared against final asthma diagnosis. Data are presented for participants with FeNO >=25ppb to <=50ppb who either did not smoke previously or are current smokers.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 11
participants
  No Previous Smoker | 11
  Current Smoker | 0

21. Primary Outcome: FeNO Values by Smoking Status: FeNO >= 50ppb
Description: Fractional Exhaled Nitric Oxide (FeNO) measurements were performed according to the "Perform FeNO Measurement" guidelines on page 7 of the NIOX MINO® User Manual (February, 2011). Methacholine Challenge (MCC) tests were performed according to the ATS guidelines and the Allergy and Asthma Specialists Procedure for conducting MCC tests. Values from the two tests were compared against final asthma diagnosis. Data are presented for participants with FeNO >=50ppb who either did not smoke previously or are current smokers.
Time Frame: approximately 1-hour
Measure: Number; unit: participants
Arm/Group | FeNO
Number analyzed (Participants) | 1
participants
  No Previous Smoker | 0
  Current Smoker | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Each subject from the time of consent until study completion.
Arm/Group | FeNO
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less